CLINICAL TRIAL: NCT00892073
Title: Combined Diazoxide and Metformin Therapy in Children With Hypothalamic Obesity Secondary to Craniopharyngioma: A Pilot Study
Brief Title: Hypothalamic Obesity Following Craniopharyngioma Surgery: A Pilot Trial of Combined Metformin and Diazoxide Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Staff Endocrinologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000008879; 9427-H1117-120C
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Hypothalamic Obesity
Keywords: Craniopharyngioma surgery; Hypothalamic Obesity; Children; Combined Diazoxide and Metformin
MeSH Terms: conditions — Sexual Infantilism | interventions — Diazoxide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diazoxide and Metformin Therapy (Experimental)
  Interventions: Drug: Diazoxide; Drug: Metformin

INTERVENTIONS:
Drug: Diazoxide — Diazoxide will be initiated at half the dose (100 mg per day) for 2 weeks to allow the insulin sensitizing action of metformin to take effect. Dosage will be increased to 200mg daily, divided twice daily with meals for 6 months.
  Other Names: Proglycem
Drug: Metformin — Metformin will be initiated at 500 mg twice daily and increased to 1000 mg twice daily over a one week period to minimize gastrointestinal side effects. the 2000mg is to be taken with meals for 6 months.
  Other Names: Novo-metformin

SUMMARY:
To study the effect of combined diazoxide-metformin therapy on body weight in youth with hypothalamic obesity following treatment for craniopharyngioma. A secondary objective is to evaluate changes in insulin resistance (IR), beta-cell function, features of the metabolic syndrome, muscle metabolism and intramyocellular lipid.

Hypothesis: Treatment with diazoxide and metformin will result in weight loss or slowed weight gain and improved metabolic profile, compared to pretreatment levels.

DETAILED DESCRIPTION:
46 children under the age of 22 years have been treated surgically for craniopharyngioma tumor and are currently followed at the Hospital for Sick Children, Toronto. Approximately 50% are obese (BMI ≥ 95th percentile for age and gender assessed from the updated Centre for Disease Control growth charts), all of whom have panhypopituitarism requiring hormone replacement therapy. These children are assessed regularly in Endocrine Clinic and also are invited to attend a comprehensive care clinic for evaluation by an endocrinologist (Principal Investigator), neurosurgical clinical nurse practitioner, dietitian, exercise physiologist, psychologist and social worker to provide multi-disciplinary dietary and exercise consultation and psychological counseling for weight related concerns. This clinic will provide the infrastructure for recruitment and follow-up of study patients. Recruitment of eight subjects for this pilot study will occur over 6 months from patients attending the comprehensive clinic. This number was chosen as it is equivalent to the number chosen in the pilot study of octreotide by Lustig which showed beneficial changes in body mass index with treatment.

This study evaluates a novel combination therapy in children with hypothalamic obesity at very high risk for complications. Evaluation of insulin resistance and metabolic changes on therapy will allow a better understanding of how insulin secretion relates to weight gain in this population. Successful therapy in a pilot setting will provide necessary data for a larger randomized trial in individuals with hypothalamic obesity including children with craniopharyngioma and others with damage to the hypothalamus secondary to other tumors, surgery or cranial irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Craniopharyngioma at least one year following surgery
* Evidence of at least one other endocrinopathy of hypothalamic origin
* Stable hormone replacement therapy (with one or more of thyroxine hydrocortisone, DDAVP, sex steroids and GH)
* Obesity, defined as weight >120% Ideal Body Weight (IBW) or BMI > 27 kg/m2, with normal weight for height before tumour diagnosis and weight gain >2SD above mean for age for 1 year following tumour treatment (41).
* Age 9 -22 years
* Minimum of 6 months of standard diet and exercise intervention (run-in period). This was chosen to allow a period of prospective measurements to establish individual baseline slope of change in BMI SDS prior to initiation of active treatment with diazoxide and metformin.

Exclusion Criteria:

* Contraindications for Metformin or Diazoxide use (history or evidence of cardiac, renal, or progressive hepatic disease , diabetes or hypoxic conditions)
* Pharmacologic doses of glucocorticoids or use of other medications known to affect glucose metabolism (e.g. beta-blockers, oral hypoglycemics)
* Growth hormone (GH) initiation in the preceding 6 months or planned initiation in the next 6 months (to rule out potential confounding effect of GH on weight / body composition and glucose metabolism).
* Use of other weight loss medications
* Inability of the family and/or patient to comply with study protocol
* Non English speaking

Ages: 9 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in BMI and BMI SDS (calculated using for Disease Control formula - www.cdc.gov.doc) over 6 months of treatment compared to change in BMI and BMI SDS over 6 month 'run-in' period (prior to study start) | 6 months prior to baseline, Baseline, 6 months after baseline

SECONDARY OUTCOMES:
Insulin secretion | Baseline to 6 months
Insulin resistance | Baseline to 6 months
Lipid profile | Baseline to 6 months
Adiponectin | Baseline to 6 months
Leptin | Baseline to 6 months
Features of the metabolic syndrome | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada